CLINICAL TRIAL: NCT06605781
Title: Enhancing Auditory Hallucination Assessment and Intervention Skills of Psychiatric Nursing Student Through AR/VR Technology and OSCE in Virtual Clinical Environments
Brief Title: Enhancing Psychiatric Nursing Skills in Auditory Hallucination Assessment Via AR/VR and Virtual OSCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NYCU113035AEF
Record Dates: First submitted 2024-08-19; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Randomized Controlled Trial
Keywords: duditory hallucination assessment; nurse student; AR/VR

STUDY DESIGN:
Intervention Model Description: The participants will be divided into experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive AR/VR technology-based group training within a virtual clinical environment during their practicum
  Interventions: Behavioral: AR/VR technology-based training
- Control group (Active Comparator): The control group will watch educational videos and participate in a general discussion group focused on auditory hallucinations.
  Interventions: Behavioral: traditional vedio and discussion group

INTERVENTIONS:
Behavioral: AR/VR technology-based training — Students will receive AR/VR Technology and OSCE in a Virtual Clinical Environment to learn how to assess and manage patients with auditory hallucination. The course was designed as a diverse and interactive learning experience, integrating a virtual clinical environment for auditory hallucinations with the application of Objective Structured Clinical Examination (OSCE). The practicum lasts approximately 15 days, with 8 hours per day. The teaching activities of the course will be held 5 times on days 4, 6, 8, 10, and 12 of the practicum. Additionally, students will have access to the AR/VR materials for self-practice during the practicum.
  Arms: Experimental group
Behavioral: traditional vedio and discussion group — Students will receive a traditional course on auditory hallucination assessment, which includes watching educational videos and participating in a general discussion group on auditory hallucinations. The practicum lasts approximately 15 days, with 8 hours per day. The teaching activities of the traditional course will be held 5 times on days 4, 6, 8, 10, and 12 of the practicum.
  Arms: Control group

SUMMARY:
The purpose of this study is to develop and evaluate AI-based virtual reality teaching resources aimed at enhancing nursing students' competencies in assessing, communicating with, and managing patients experiencing auditory hallucinations. Specifically, this study seeks to improve the ability of nursing students to effectively assess auditory hallucinations, facilitate better communication with patients experiencing such disturbances, and strengthen their skills in managing these symptoms through the implementation of virtual reality-based educational scenarios.

DETAILED DESCRIPTION:
This study employs a quasi-experimental design and uses a convenience sampling method to select senior students from a university nursing program as participants. The study aims to recruit 150 nursing students. The research involves two institutions, with participants being divided into groups within each institution. The students will be randomly assigned by computer into two groups: an experimental group and a control group. The experimental group will receive AR/VR technology-based group training within a virtual clinical environment during their practicum, while the control group will watch educational videos and participate in a general discussion group focused on auditory hallucinations.

Data will be collected using Google Forms at two time points: baseline and post-intervention. The research instruments include:

1. A self-assessment questionnaire on confidence in auditory hallucination assessment and intervention;
2. A scale measuring nursing students' knowledge, attitudes, and perceived empathy toward auditory hallucinations;
3. The Auditory Hallucination Situational Involvement and Empathy Scale;
4. An OSCE (Objective Structured Clinical Examination) evaluation form that assesses auditory hallucination assessment skills, empathy toward auditory hallucinations, communication skills, and the ability to manage auditory hallucinations." Data will be analyzed using IBM SPSS 24.0 for descriptive statistics and for comparing outcomes between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students who are about to undertake their psychiatry practicum.
* Those who are willing to join the study and sign the consent form.
* Those who are willing to bring a smartphone to connect with VR360 and watch the video.
* Those who are willing to use their smartphone for research purposes (a smartphone will be provided by the research team if needed).

Exclusion Criteria:

* Individuals with hearing or vision impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Auditory Hallucination Situational Involvement and Empathy | at baseline on day 2 or 3 of the 15-day practicum (T0) and on day 15 of the practicum, three days after the intervention has finished (T1)
  To assess the impact of the intervention on empathy, Schutte and Stilinović's (2017) method was used, employing the Situational Scale of Empathetic Responses (SSER) with 15 items. These are divided into two categories: ① Empathic Perspective Taking (7 items) and ② Empathic Concern (8 items). Participants imagined interacting with a person hearing voices and rated the items on a 5-point Likert scale, from 'strongly disagree' (1) to 'strongly agree' (5). Higher scores indicate greater empathy in auditory hallucination scenarios.
OSCE Evaluation Form for Auditory Hallucination Assessment and Intervention | at baseline on day 2 or 3 of the 15-day practicum (T0) and on day 15 of the practicum, three days after the intervention has finished (T1)
  This form is part of the "Application of AR/VR Technology and OSCE in a Virtual Clinical Environment" teaching practice project. Both the experimental and control groups will watch videos; however, the control group will watch standard videos, while the experimental group will use AR/VR technology within a virtual clinical environment. Both groups will be assessed using OSCE combined with the virtual clinical environment.
  The evaluation form, developed by the researcher, will undergo content validity review by experts once the videos are completed. Different versions of the virtual clinical environment and OSCE assessment will be used before and after the intervention. The study plans to develop four different versions, all of which will be reviewed by experts and piloted.
Self-Assessment Questionnaire on Confidence in Auditory Hallucination Assessment and Intervention | at baseline on day 2 or 3 of the 15-day practicum (T0) and on day 15 of the practicum, three days after the intervention has finished (T1)
  This section consists of a self-designed questionnaire by the researcher, primarily aimed at measuring students' confidence levels before and after the implementation of the teaching intervention. It includes 7 items and serves as a simple assessment tool.
Nursing Students' Knowledge, Attitudes, and Perceived Empathy Toward Auditory Hallucinations | at baseline on day 2 or 3 of the 15-day practicum (T0) and on day 15 of the practicum, three days after the intervention has finished (T1)
  This assessment tool, developed by Mawson (2014), consists of 11 items related to statements about knowledge, attitudes, and empathy toward auditory hallucinations. Nursing students are asked to respond to these statements using a 5-point Likert scale, with responses ranging from "strongly agree" (5) to "strongly disagree" (1). These statements remain unchanged in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu Yueh Yang, PhD, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taipei City, Taiwan